CLINICAL TRIAL: NCT04034134
Title: A Phase Ⅱ Study to Evaluate the Safety and Efficacy of Jaktinib Hydrochloride Tablets in the Treatment of Severe Alopecia Areata.
Brief Title: Study to Evaluate the Safety and Efficacy ofJaktinib Hydrochloride Tablets in Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK003
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jaktinib Hydrochloride Tablets 50mg bid (Experimental): Oral tablet for 24 weeks
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Jaktinib Hydrochloride Tablets 150mg qd (Experimental): Oral tablet for 24 weeks
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Jaktinib Hydrochloride Tablets 200mg qd (Experimental): Oral tablet for 24 weeks
  Interventions: Drug: Jaktinib Hydrochloride Tablets

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — 50 mg twice-daily (BID)
  Arms: Jaktinib Hydrochloride Tablets 50mg bid
Drug: Jaktinib Hydrochloride Tablets — 150 mg quaque die (QD)
  Arms: Jaktinib Hydrochloride Tablets 150mg qd
Drug: Jaktinib Hydrochloride Tablets — 200 mg quaque die (QD)
  Arms: Jaktinib Hydrochloride Tablets 200mg qd

SUMMARY:
This was an open-label, Multi-center, randomized phase Ⅱ study. Patients with severe Alopecia Areata were randomized to receive 50mg bid, 150mg qd or 200 mg qd of oral Jaktinib Hydrochloride Tablets.

ELIGIBILITY:
Inclusion Criteria:

* 18 years age or older ,male or female；
* Alopecia areata diagnosed clinically；
* Patients with alopecia accounting for 50% or more of the total scalp area and stable for at least 6 months or more；
* Patients can complete treatment for at least six months；
* Requirements for pregnant or lactating female and male and female of childbearing age；Female patients must be satisfied：Menopause (defined as no menstruation for at least one year);Or have been surgically sterilized；Or have fertility, but must satisfy：Pregnancy tests conducted within 7 days before randomization must be negative；And agree to use appropriate contraceptive methods throughout the trial period, including at least one barrier method；And no breastfeeding；Male patients must agree to use appropriate contraceptive measures throughout the trial, including at least one barrier method；
* Patients are voluntarily enrolled in the Study and can be treated and visited according to the requirements of the protocol after signing the Informed Consent Form；

Exclusion Criteria:

* Alopecia caused by syphilitic alopecia, thyroid disease, trichotilomania, head moss, connective tissue disease, infection, zinc deficiency and iron deficiency;
* Patients with acute diffuse alopecia areata (ADTAFS)
* Patients with active tuberculosis
* The following diseases were combined within 6 months before randomization:thyroid diseases ，liver diseases, malnutrition, heart diseases, nervous system diseases, gastrointestinal disorders, tumors and psychiatric diseases
* HIV positive, active hepatitis B virus positive (HBsAg or HBeAg positive) and HCV-RNA positive at screening；
* Other patients with abnormal history or clinical manifestations that may affect participants participation in the study or may confuse the results of the study；
* Within two weeks before randomization，Patients who received glucocorticoid topical therapy, anthracene ointment, minoxidil, SADBE/DPCP contact immunotherapy, photochemotherapy or cryotherapy；
* Before randomization，oral or injected any medicines to treat hair loss (including the glucocorticoids was detected in injection, systemic corticosteroids, antihistamines, stephania drugs, glycyrrhizin, glycine, methionine compound tablet, compound glycyrrhizin glucoside) and other liquorice extract, ring spore element, anti TNF antibody, IFN - gamma, IL - 2 antibodies, for alopecia areata therapy of traditional Chinese medicine and other JAK inhibitor) and washout period less than seven half-life of patients;
* Participants in a clinical trial of any drug or medical device within 4 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Effective rate | From randomization of the first subject until the last subject complete 6 months treatment
  Effective rate = (cure + obvious effect + effective)/total cases *100%;

SECONDARY OUTCOMES:
SALT score change | From randomization of the first subject until the last subject complete 6 months treatment
  Score and take photos (4 areas on the head), taking photos in the same position and light condition each time;
Quality of Life (AASIS) | From randomization of the first subject until the last subject complete 6 months treatment
  AASIS was used to score the quality of life of the subjects

OTHER OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | From randomization of the first subject until the last subject complete 6 months treatment
  Patients with adverse events/all patients *100%

CONTACTS AND LOCATIONS:
Overall Officials: qianjin Lu, MD, Principal Investigator — Central South University
Locations (2):
- China (2):
  - Chongqing Chinese Traditional Medicine Hospital, Chongqing, Chongqing Municipality
  - The second xaingya hospital of central south university, Changsha, Hunan